CLINICAL TRIAL: NCT01696201
Title: Effect of a Supervised Exercise Program During Whole Pregnancy on Outcomes and Level of Depression. A Randomized Controlled Trial
Brief Title: Effect of Physical Exercise Program on Outcomes and Level of Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Madrid (Other)
Responsible Party: Principal Investigator, María Perales Santaella, PhD student, Technical University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pregnancy outcomes
Record Dates: First submitted 2012-09-17; First posted 2012-09-28 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2012-09

CONDITIONS: Pregnancy
Keywords: Pregnancy, outcomes, depression, mood, physical exercise
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention): Sedentary pregnant women
- Exercise group (Experimental): Exercise program
  Interventions: Behavioral: Exercise group

INTERVENTIONS:
Behavioral: Exercise group — Supervised physical conditioning program of three 55-60 minute sessions per week during whole pregnancy (from week 9 to 38). Each session consists of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvic floor muscles training.
  Aerobic activity was prescribed at light to moderate intensity, aiming for 55-60 of maximal heart rate. All subjects wore a heart rate (HR) monitor (Polar FT7) during the training sessions to ensure that exercise intensity was light to moderate.
  Arms: Exercise group

SUMMARY:
Due to physical and physiological changes that occur in pregnant women, depression is very common during this period. Recent research findings indicate that antenatal maternal mood state impacts on babies health. Nowadays, many researchers are focussed on examining the effects of physical exercise on foetal and maternal outcomes.

The main aim of this study was to assess the effectiveness of a supervised exercise program consisted of 25-30 minutes of cardiovascular exercise,10 minutes of specific exercises (strength and balance exercises), and 10 minutes of pelvis floor muscles training, on the prevention and treatment of depression in pregnant women. Additionally, the other purpose of the study was to analyze the effects of depression and physical exercise on outcomes.

Hypothesis: Pregnant women who do regular exercise during their pregnancies would have a better mood state than pregnant women who are sedentary, without having any negative effect on outcomes.

DETAILED DESCRIPTION:
BACKROUND: Recent studies have estimated the prevalence of depression during pregnancy at between 10% and 30%. This state can produce negative effects on the fetus as:

* Affect cerebral development
* Increase the risk of preterm birth and low birth weight
* Increase the risk of childhood overweight problems
* Adverse impact on the cognitive, emotional, social, and behavioural development of infants

Due to the possible side effect of antidepressants on mother and fetus, its necessary to examine alternative solutions to this state.

ELIGIBILITY:
Inclusion Criteria:

* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines
* Being able to communicate in spanish
* Giving birth at Hospital Universitario de Fuenlabrada

Exclusion Criteria:

* Multiparity
* Obstetrician complications
* Being interested in the study after 18 weeks
* Not being regular in physical exercise program
* Younger than 18 years old

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change from level of depression at the end of the pregnancy | Up to 36 weeks
  The Center for Epidemiological Studies-Depression scale (CES-D) was administered to all pregnant women at the beginning and at the end of their pregnancies

SECONDARY OUTCOMES:
Maternal outcome | Time spending in each stages of labor
  Time of stages of labor (min)
Fetal outcome | 1-5 minutes after labor
  Apgar score

OTHER OUTCOMES:
Maternal outcome | Between 12 and 38 weeks
  Constipation (yes/not)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Barakat, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politecnica de Madrid, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735